CLINICAL TRIAL: NCT03704168
Title: Safety and Efficacy of Cryoablation in Management of Sialorrhea in Patients With Neurological Disorders.
Acronym: SECAMS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never launched.
Sponsor: Dean Nakamoto (Other)
Responsible Party: Sponsor-Investigator, Dean Nakamoto, Division Chief, Abdominal Imaging - UH Cleveland Medical Center, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SECAMS
Record Dates: First submitted 2018-02-23; First posted 2018-10-12 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Sialorrhea; Neurologic Disorder
MeSH Terms: conditions — Sialorrhea; Nervous System Diseases | interventions — Cryosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CRYOABLATION ARM (Experimental)
  Interventions: Device: CRYOABLATION

INTERVENTIONS:
Device: CRYOABLATION — The SeedNet® System induces freezing and thawing at the tip of the needle. These freezing and thawing processes are based on the Joule-Thomson effect. The unique technology of the SeedNet® System provides extremely rapid freeze and thaw operations. The system's software controls the flow of gases from the gas sources, through the manifold, to the needle and probe tips. The system can immediately switch from the freezing process to the thawing process, after which the needle can be released. This device is an FDA-cleared medical device. This IDE application is to allow for use of the commercially available device in a new clinical indication, namely cryoablation of the submandibular glands.
  Other Names: SeedNet® System

SUMMARY:
To evaluate safety of cryoablation of submandibular glands in management of sialorrhea in neurologically impaired populations.

Secondary Objective: To evaluate efficacy of cryoablation of submandibular glands in management of sialorrhea in neurologically impaired populations.

Duration:

Estimation for Recruitment: 12 months Estimation for Procedure/Trial: 1 visit with an overnight observation Estimation for Subject Follow Up: 7 days, 14 days, 28 days, 90 days, and 180 days, post ablation, with ultrasound of the bilateral submandibular glands at 28 days and 180 days post ablation Total Expected Duration for Clinical Trial: 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and assent (as appropriate) obtained from the subject/caregiver who opted voluntarily to participate in the procedure
2. Male or female 2 to 65 years of age
3. Confirmed diagnosis of sialorrhea as documented in their medical record
4. Clinically stable with no significant changes in health status in the 2 weeks before the ablation
5. Patients diagnosed with cerebral palsy, or other neurological impairment documented in their medical record

Exclusion Criteria:

1. Open sores/ulcers on skin overlying the submandibular glands
2. Contraindications to surgery/general anesthesia e.g; coagulopathies, life threatening arrhythmias
3. Upper respiratory airway obstruction, e.g: severe dystonia
4. History of previous local surgery
5. Any congenital abnormalities that may preclude cryoablation, such as vascular abnormalities or atypical size/location
6. Patients that have received salivary gland Botulinum toxin injections within the prior 3 months
7. Subjects unlikely to complete the study as determined by the principle investigator

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety of cryoablation of submandibular glands in management of sialorrhea in neurologically impaired populations. | 2 years
  1. Safety Parameters: Major adverse events will be submitted to the Agency and be reviewed by the medical monitor. In case unexpected events should occur we will evaluate and report them.
  2 Methods for Analyzing Safety Parameters: Prior to the enrollment of the first research subject, the study sponsor will organize and conduct an initial meeting for the medical monitor. The medical monitor will review AE logs, deviation logs, procedural details, call logs, phone scripts, study progress notes, patient medical charts, and completed questionnaires, every 5 patients, or quarterly, whichever takes place first. The sponsor-investigator will oversee the conduct of the medical monitor. Directives provided by the medical monitor will be reported accordingly and as necessary to the Food and Drug Administration and the IRB.

SECONDARY OUTCOMES:
To evaluate efficacy of cryoablation of submandibular glands in management of sialorrhea in neurologically impaired populations. | 2 years
  1. Efficacy Parameters:
     Efficacy is defined as reduced score on the Drooling Impact Scale (range: 10-100) at baseline, 1 and 6 months interval with-in subject self-assessment.
  2. Methods for Analyzing Efficacy Parameters:
  We will qualitatively assess the impact of drooling on patients, their families, and/or caretakers, at baseline, then twice post procedurally, using a questionnaire. The questionnaire known as the Drooling Impact Scale 'DIS' has been devised to evaluate longitudinal changes in children with neurological disorders, and quantify short- to medium-term treatment benefits of saliva-control interventions.